CLINICAL TRIAL: NCT03018418
Title: A Prospective Pilot Study to Evaluate the Feasibility of Intensity Modulated Proton Therapy in Reducing Toxicity in Anal Cancer
Brief Title: Proton Therapy in Reducing Toxicity in Anal Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jordan Kharofa (Other)
Responsible Party: Sponsor-Investigator, Jordan Kharofa, Assistant Professor, University of Cincinnati
Organization: University of Cincinnati (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCCI-GI-16-01
Record Dates: First submitted 2017-01-10; First posted 2017-01-12 (Estimated); Results first posted 2023-10-05 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Anus Neoplasms
Keywords: Anal Cancer
MeSH Terms: conditions — Anus Neoplasms | interventions — Proton Therapy; Drug Therapy; Fluorouracil; Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Proton Therapy and Chemotherapy (Experimental): Standard chemoradiation using 5-FU, Mitomycin, with pencil beam proton radiotherapy
  Interventions: Radiation: Proton therapy; Drug: Chemotherapy

INTERVENTIONS:
Radiation: Proton therapy — Primary target volume 50.4-54 CGE in 28-30 fractions; Nodal volumes 42-54 CGE in 28-30 fractions
Drug: Chemotherapy — 5FU 1000 mg/m2/day as 96 hour infusion days 1-5 and 29-33; Mitomycin 10mg/m2 days 1 and 29
  Other Names: 5FU; Mitomycin

SUMMARY:
The purpose of this research study is to determine whether the amount of radiation given to the normal areas around the anal cancer can be reduced by using Proton Therapy while reducing the side effects that are seen with standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* Karnofsky Performance Status >70%
* Histologically documented squamous or basaloid carcinoma of the anal canal
* Stage T2-4 disease with any N category

Exclusion Criteria:

• Patients with a life expectancy of < 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-01-04 (Actual); Primary Completion 2022-04-07 (Actual); Study Completion 2025-07-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Kharofa, MD, Principal Investigator — University of Cincinnati
Locations (1):
- UC Health, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Stage II and III Anal Cancer: Patients with histologically confirmed squamous or basaloid carcinoma of the anal canal were eligible if they were at least 18 years old with a Karnofsky performance status > 70%, AJCC eighth edition cT2-4 disease with any N category, life expectancy >3 months, and acceptable organ and bone marrow function. Women who were not postmenopausal had to have a negative urine or serum pregnancy test. History and physical examination (including anal and groin evaluation) had to be performed within 21 days of trial registration.
Period: Overall Study
Arm/Group | Patients With Stage II and III Anal Cancer
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Proton Therapy and Chemotherapy
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 4
Age, Continuous [Median (Full Range); unit: years] | 56 [31 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Rates of Acute Toxicity
Description: Grade 3 or greater hematologic, gastrointestinal, genitourinary, and dermatologic toxicity
Time Frame: 3 months
Population: The population is the subjects that had at least one adverse event that was grade 3 or higher in one of the following categories: hematologic, gastrointestinal, genitourinary, and dermatologic
Measure: Count of Participants; unit: Participants
Groups:
- Grade 3+ Hematologic, Gastrointestinal, Genitourinary, and Dermatologic Toxicity: Subjects with grade 3+ Adverse events that fall within the following categories: hematologic, gastrointestinal, genitourinary, and dermatologic
Arm/Group | Grade 3+ Hematologic, Gastrointestinal, Genitourinary, and Dermatologic Toxicity
Number analyzed (Participants) | 14
Participants | 12

2. Secondary Outcome: Rates of Late Toxicity
Description: Grade 3 or greater hematologic, gastrointestinal, genitourinary, and dermatologic toxicity
Time Frame: every 6 months up to 60 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Grade 3+ Hematologic, Gastrointestinal, Genitourinary, and Dermatologic Toxicity
Number analyzed (Participants) | 14
Participants | 6

3. Secondary Outcome: Complete Response Rate
Description: Complete response was clinically determined by digital rectal examination and proctosigmoidoscopy supplemented with pelvic axial imaging. Biopsy was not required. The complete response was the absence of disease based on these evaluations. Any measurable disease at 6 months from the completion of chemoradiation will be considered a local treatment failure. Any tumor recurrence in the anus in patients who initially had a complete response will be considered a local recurrence.
Time Frame: at 6 months from the completion of chemoradiation
Measure: Count of Participants; unit: Participants
Groups:
- Subjects With Complete Response Rate: 14 represents the total sample size of the study. 11 met complete clinical response at 6 months.
Arm/Group | Subjects With Complete Response Rate
Number analyzed (Participants) | 14
Participants | 11

4. Secondary Outcome: Local Progression Free Survival
Description: This is the percentage of subjects that were free of local progression.
Time Frame: every 6 months up to 60 months
Measure: Count of Participants; unit: Participants
Groups:
- Local Progression Free Survival for 14 Subjects: This is the local progression free survival for 14 subjects.
Arm/Group | Local Progression Free Survival for 14 Subjects
Number analyzed (Participants) | 14
Participants | 12

5. Secondary Outcome: Overall Survival
Description: This is an estimated percentage of participants that is alive at 2 years.
Time Frame: every 6 months up to 24 months
Population: time from the date of registration to the date of death due to all causes
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Groups:
- Overall Survival for 14 Subjects: time from the date of registration to the date of death due to all causes
Arm/Group | Overall Survival for 14 Subjects
Number analyzed (Participants) | 14
percentage of subjects | 76 [73 to 92]

6. Secondary Outcome: Distant Metastases Free Survival
Description: This is the percentage of subjects that were free of distant metastases.
Time Frame: every 6 months up to 60 months
Measure: Count of Participants; unit: Participants
Groups:
- Distant Metastases Free Survival for 14 Subjects: Distant metastases free survival for 14 subjects
Arm/Group | Distant Metastases Free Survival for 14 Subjects
Number analyzed (Participants) | 14
Participants | 13

7. Secondary Outcome: Quality of Life Changes
Description: Utilization of the Patient Reported Outcomes- Common Toxicity Criteria for Adverse Events at pretreatment and up to 12 months. This measure used the difference total score for each subject's baseline and latest PROCTCAE available. The reported statistic is the number of subjects that showed a reduction in scores between the two time points.
Time Frame: before treatment and 12 months after start of treatment
Population: This measure examines all 14 subjects.
Measure: Count of Participants; unit: Participants
Groups:
- Quality of Life Changes for 14 Subjects: Utilization of the Patient Reported Outcomes- Common Toxicity Criteria for Adverse Events at pretreatment, 2 weeks, 4 weeks, 3, 6, and 12 months
Arm/Group | Quality of Life Changes for 14 Subjects
Number analyzed (Participants) | 14
Participants | 9

ADVERSE EVENTS:
Time Frame: AEs were collected from the start of treatment to 90 days after post treatment. If an AE was one of the subset of AEs listed below, then the AE was tracked beyond 90 days until resolution or the end of the study (60 months). The subset of AEs are: (1) AEs that may be reasonably related to the organ systems within the study treatment field (such as the GI/GU/Vaginal/Skin/pelvic bone organ systems) and (2) all SAEs.
Description: The definition does not differ from clinicaltrials.gov.
Groups:
- Adverse Events for All 14 Subjects: This is a summary of adverse events for all 14 subjects in the study.
Arm/Group | Adverse Events for All 14 Subjects
All-Cause Mortality (participants affected / at risk) | 2/14
Serious Adverse Events (participants affected / at risk) | 7/14
Other Adverse Events (participants affected / at risk) | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adverse Events for All 14 Subjects (N=14)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1) — Cardiac Pain-unspecified
Cardiac disorders - Other, specify (Cardiac disorders) | 2 (2) — NSTEMI - type 1
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (3) — Pneumonia
Infections and infestations - Other, specify (Infections and infestations) | 1 (2) — E. Coli Sepsis
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1) — Failure to Thrive
Pregnancy, puerperium and perinatal conditions - Other, specify (Pregnancy, puerperium and perinatal conditions) | 1 (1) — Placenta Increta
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (1) — Altered Mental Status
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (5) — Acute Exacerbation of COPD
Respiratory, thoracic and mediastinal disorders - Other, specify (Reproductive system and breast disorders) | 1 (4) — Acute on chronic Hypoxic and Hypercarbic Respiratory Failure
Urinary tract infection (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adverse Events for All 14 Subjects (N=14)
Abdominal pain (Gastrointestinal disorders) | 6 (11)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1)
Anal pain (Gastrointestinal disorders) | 8 (8)
Anemia (Blood and lymphatic system disorders) | 6 (19)
Anorexia (Metabolism and nutrition disorders) | 7 (11)
Anxiety (Psychiatric disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Burn (Injury, poisoning and procedural complications) | 2 (2)
Tachycardia (Cardiac disorders) | 3 (3)
Chills (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Creatinine increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 12 (20)
Diarrhea (Gastrointestinal disorders) | 10 (18)
Dizziness (Nervous system disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 5 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Edema limbs (General disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (General disorders) | 9 (9)
Fecal incontinence (Gastrointestinal disorders) | 3 (3)
Fever (General disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 6 (10)
Floaters (Eye disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) — Stinging sensation in anal region
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) — Rectal Cramping
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) — dark red mucous small clot in stool
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (4)
Headache (Nervous system disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (3)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Immune system disorders - Other, specify (Immune system disorders) | 1 (1) — Neutropenic Fever
Infections and infestations - Other, specify (Infections and infestations) | 1 (2) — E. Coli Sepsis
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) — C. Diff
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) — Hospital Acquired Pneumonia
Insomnia (Psychiatric disorders) | 1 (1)
Localized edema (General disorders) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 9 (35)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1) — Failure to Thrive
Mucositis oral (Gastrointestinal disorders) | 5 (7)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 10 (19)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) — Sciatica
Neutrophil count decreased (Investigations) | 6 (9)
Non-cardiac chest pain (General disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 2 (4)
Pain (General disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Paresthesia (Nervous system disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Platelet count decreased (Investigations) | 9 (15)
Proctitis (Gastrointestinal disorders) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 2 (2)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1) — Urinary Hesitancy
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1) — Nocturia
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1) — Weak Stream
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Acute Respiratory Failure
Sinus tachycardia (Cardiac disorders) | 2 (2)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) — Erythema on face from 5FU
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) — Perianal Skin Irritation
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) — Perianal Skin Pain
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (3)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Superficial soft tissue fibrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 8 (10)
Urinary incontinence (Renal and urinary disorders) | 5 (6)
Urinary retention (Renal and urinary disorders) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2)
Urinary tract pain (Renal and urinary disorders) | 4 (7)
Urinary urgency (Renal and urinary disorders) | 5 (6)
Urine discoloration (Renal and urinary disorders) | 5 (5)
Vaginal discharge (Reproductive system and breast disorders) | 2 (2)
Vaginal dryness (Reproductive system and breast disorders) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (7)
Weight gain (Investigations) | 1 (1)
Weight loss (Investigations) | 2 (2)
White blood cell decreased (Investigations) | 10 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-31): https://cdn.clinicaltrials.gov/large-docs/18/NCT03018418/Prot_SAP_000.pdf